CLINICAL TRIAL: NCT03045887
Title: A Single-centre, Double-blind (Sponsor Open), Placebo Controlled Two Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of GSK2292767 as a Dry Powder in Healthy Participants Who Smoke Cigarettes
Brief Title: Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of GSK2292767 in Healthy Participants Who Smoke Cigarettes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202062; 2016-003188-21 (EudraCT Number)
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: repeat dose; GSK2292767; smoke; tolerability; safety; dry powder inhalation; pharmacokinetics; single dose
MeSH Terms: conditions — Asthma | interventions — GSK2292767

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part A Cohort 1: Placebo- GSK2292767 (GSK) 200 µg-GSK 1000 µg (Experimental): Subjects will receive an inhaled single dose of placebo in Period 1, GSK2292767 200 µg in Period 2, and GSK2292767 1000 µg in Period 3. There will be a washout of approximately 4 weeks between doses.
  Interventions: Drug: GSK2292767 50 μg; Drug: GSK2292767 500 μg; Drug: Placebo
- Part A Cohort 1: GSK 50 µg-Placebo-GSK 1000 µg (Experimental): Subjects will receive an inhaled single dose of GSK2292767 50 µg in Period 1, placebo in Period 2, and GSK2292767 1000 µg in Period 3. There will be a washout of approximately 4 weeks between doses.
  Interventions: Drug: GSK2292767 50 μg; Drug: GSK2292767 500 μg; Drug: Placebo
- Part A Cohort 1: GSK 50 µg- GSK 200 µg-Placebo (Experimental): Subjects will receive an inhaled single dose of GSK2292767 50 µg in Period 1, GSK2292767 200 µg in Period 2, and placebo in Period 3. There will be a washout of approximately 4 weeks between doses.
  Interventions: Drug: GSK2292767 50 μg; Drug: Placebo
- Part A Cohort 1: GSK 50 µg-GSK 200 µg-GSK 1000 µg (Experimental): Subjects will receive an inhaled single dose of GSK2292767 50 µg in Period 1, GSK2292767 200 µg in Period 2, and GSK2292767 1000 µg in Period 3. There will be a washout of approximately 4 weeks between doses.
  Interventions: Drug: GSK2292767 50 μg; Drug: GSK2292767 500 μg
- Part A Cohort 2: Placebo-GSK 500 µg-GSK 2000 µg (Experimental): Subjects will receive an inhaled single dose of placebo in Period 1, GSK2292767 500 µg in Period 2, and GSK2292767 2000 µg in Period 3. There will be a washout of approximately 4 weeks between doses.
  Interventions: Drug: GSK2292767 500 μg; Drug: Placebo
- Part A Cohort 2: GSK 100 µg-Placebo- GSK 2000 µg (Experimental): Subjects will receive an inhaled single dose of GSK2292767 100 µg in Period 1, placebo in Period 2, and GSK2292767 2000 µg in Period 3. There will be a washout of approximately 4 weeks between doses.
  Interventions: Drug: GSK2292767 50 μg; Drug: GSK2292767 500 μg; Drug: Placebo
- Part A Cohort 2: GSK 100 µg-GSK 500 µg-Placebo (Experimental): Subjects will receive an inhaled single dose of GSK2292767 100 µg in Period 1, GSK2292767 500 µg in Period 2 and placebo in Period 3. There will be a washout of approximately 4 weeks between doses.
  Interventions: Drug: GSK2292767 50 μg; Drug: GSK2292767 500 μg; Drug: Placebo
- Part A Cohort 2: GSK 100 µg-GSK 500 µg-GSK 2000 µg (Experimental): Subjects will receive an inhaled single dose of GSK2292767 100 µg in Period 1, GSK2292767 500 µg in Period 2, GSK2292767 2000 µg in Period 3. There will be a washout of approximately 4 weeks between doses.
  Interventions: Drug: GSK2292767 50 μg; Drug: GSK2292767 500 μg
- Part B: GSK (Experimental): Subjects will receive inhaled repeat dose of GSK2292767 2000 µg once daily for 14 days.
  Interventions: Drug: GSK2292767 500 μg
- Part B: Placebo (Experimental): Subjects will receive inhaled repeat dose of placebo once daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2292767 50 μg — GSK2292767 50 μg blended with lactose and magnesium stearate per blister as powder for inhalation
  Arms: Part A Cohort 1: GSK 50 µg- GSK 200 µg-Placebo; Part A Cohort 1: GSK 50 µg-GSK 200 µg-GSK 1000 µg; Part A Cohort 1: GSK 50 µg-Placebo-GSK 1000 µg; Part A Cohort 1: Placebo- GSK2292767 (GSK) 200 µg-GSK 1000 µg; Part A Cohort 2: GSK 100 µg-GSK 500 µg-GSK 2000 µg; Part A Cohort 2: GSK 100 µg-GSK 500 µg-Placebo; Part A Cohort 2: GSK 100 µg-Placebo- GSK 2000 µg
Drug: GSK2292767 500 μg — GSK2292767 500 μg blended with lactose and magnesium stearate per blister as powder for inhalation
  Arms: Part A Cohort 1: GSK 50 µg-GSK 200 µg-GSK 1000 µg; Part A Cohort 1: GSK 50 µg-Placebo-GSK 1000 µg; Part A Cohort 1: Placebo- GSK2292767 (GSK) 200 µg-GSK 1000 µg; Part A Cohort 2: GSK 100 µg-GSK 500 µg-GSK 2000 µg; Part A Cohort 2: GSK 100 µg-GSK 500 µg-Placebo; Part A Cohort 2: GSK 100 µg-Placebo- GSK 2000 µg; Part A Cohort 2: Placebo-GSK 500 µg-GSK 2000 µg; Part B: GSK
Drug: Placebo — Lactose as powder for inhalation
  Arms: Part A Cohort 1: GSK 50 µg- GSK 200 µg-Placebo; Part A Cohort 1: GSK 50 µg-Placebo-GSK 1000 µg; Part A Cohort 1: Placebo- GSK2292767 (GSK) 200 µg-GSK 1000 µg; Part A Cohort 2: GSK 100 µg-GSK 500 µg-Placebo; Part A Cohort 2: GSK 100 µg-Placebo- GSK 2000 µg; Part A Cohort 2: Placebo-GSK 500 µg-GSK 2000 µg; Part B: Placebo

SUMMARY:
This study is the first administration of GSK2292767 to humans. The study will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and repeat inhaled doses of GSK2292767 in healthy smokers. This study is intended to provide sufficient confidence in the safety of the molecule and preliminary information on target engagement to allow progression to further repeat dose and proof of mechanism studies. This is a two part, single site, randomized, double-blind (sponsor open), placebo controlled study. Part A will consist of two 3-period interlocking cohorts to evaluate the safety, tolerability and pharmacokinetics of ascending single doses of GSK2292767 administered as a dry powder inhalation. Part B is planned to follow Part A and progression will be based on an acceptable safety, tolerability and pharmacokinetic profiles. Subjects will receive repeat doses of GSK2292767 once daily for 14 days during Part B.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent
* Participants who are overtly healthy as determined by medical evaluation including (medical history, physical examination, laboratory tests, and cardiac monitoring). A participant with a clinical abnormality or laboratory parameters outside the reference range expected for them and the population being studied may be included only if the Investigator believes that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or outcomes
* Participants who are current daily cigarette smokers (manufactured and self-rolled). Must have smoked regularly in the 12-month period preceding the screening visit
* Normal spirometry (FEV1 >=80% of predicted) at screening
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 18 to 31 kg/square meter (m^2) (inclusive)
* Male and female

  * Male participants: A male participant must agree to use contraception as detailed in the protocol during the treatment period and for at least from the time of first dose of study medication until at least 55 (5x11) hours plus an additional 90 days after the last dose of study medication and refrain from donating sperm during this period. GSK2292767 has a predicted half-life of approximately 11 hours
  * Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential (WOCBP)
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol

Exclusion Criteria:

* History or presence of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data
* Abnormal blood pressure as determined by the investigator
* Alanine transaminase (ALT) >1.5xupper limit of normal (ULN)
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Average corrected QT interval by Fridericia's formula (QTcF) >450 milliseconds (msec) (based on triplicate ECGs)
* Participants who have asthma or a history of asthma (except in childhood and which has now remitted)
* Past or intended use of over-the-counter or prescription medication including herbal medications within 14 days prior to dosing. Specific concomitant medications listed in protocol may be allowed
* Live vaccine(s) within 1 month prior to screening, or plans to receive such vaccines during the study
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters (mL) within 56 days
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day
* Current enrolment or past participation within the last 90 days of exposure to any other clinical study involving an investigational study treatment or any other type of medical research
* Presence of Hepatitis B surface antigen (HBsAg) at screening Positive Hepatitis C antibody test result at screening
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment
* Positive pre-study drug/alcohol screen
* Positive human immunodeficiency virus (HIV) antibody test
* Regular use of known drugs of abuse
* Regular alcohol consumption within 3 months prior to the study defined as: An average weekly intake of >14 units for males and females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study
* Participants who are unable to produce a total weight of at least 100 milligrams (mg) of selected sputum during sputum induction at screening
* Participants whose primary consumption of tobacco is via methods other than cigarettes (manufactured or self-rolled). Primary methods of tobacco consumption that are excluded include, but are not limited to pipes and cigars

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=202062

REFERENCES:
- [Background] Begg M, Edwards CD, Hamblin JN, Pefani E, Wilson R, Gilbert J, Vitulli G, Mallett D, Morrell J, Hingle MI, Uddin S, Ehtesham F, Marotti M, Harrell A, Newman CF, Fernando D, Clark J, Cahn A, Hessel EM. Translation of Inhaled Drug Optimization Strategies into Clinical Pharmacokinetics and Pharmacodynamics Using GSK2292767A, a Novel Inhaled Phosphoinositide 3-Kinase delta Inhibitor. J Pharmacol Exp Ther. 2019 Jun;369(3):443-453. doi: 10.1124/jpet.119.257311. Epub 2019 Apr 2. PMID 30940692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a two part, single site, randomized, double-blind (sponsor open), placebo controlled study in healthy smokers. Study was conducted in the United Kingdom.
Pre-assignment Details: Part A comprised of two cohorts, each of which consisted of 3 treatment periods with 4 treatment sequences. Out of 98 screened participants, 37 were randomized, 58 were screen failures and 3 were retained as reserve participants. In Part B, 12 participants were included, 11 of them were taken from Part A and 1 additional participant only for Part B
Groups:
- Part A: Placebo/200 µg GSK2292767/1000 µg GSK2292767: Part A consisted of two cohorts each containing three treatment periods with four treatment sequences. Participants randomized to Sequence 1 were administered a single dose of placebo in Period 1, 200 µg GSK2292767 in Period 2 and 1000 µg GSK2292767 in Period 3. The treatment was administered via ELLIPTA Dry Powder Inhaler (DPI). There was a period of 4 weeks between doses for an individual participant.
- Part A:50 µg GSK2292767/Placebo/1000 µg GSK2292767: Part A consisted of two cohorts each containing three treatment periods with four treatment sequences. Participants randomized to Sequence 2 were administered a single dose of 50 µg GSK2292767 in Period 1, placebo in Period 2 and 1000 µg GSK2292767 in Period 3. The treatment was administered via ELLIPTA DPI. There was a period of 4 weeks between doses for an individual participant.
- Part A:50 µg GSK2292767/200 µg GSK2292767/Placebo: Part A consisted of two cohorts each containing three treatment periods with four treatment sequences. Participants randomized to Sequence 3 were administered a single dose of 50 µg GSK2292767 in Period 1, 200 µg GSK2292767 in Period 2 and placebo in Period 3. The treatment was administered via ELLIPTA DPI. There was a period of 4 weeks between doses for an individual participant.
- Part A:50 µg GSK2292767/200 µg GSK2292767/1000 µg GSK2292767: Part A consisted of two cohorts each containing three treatment periods with four treatment sequences. Participants randomized to Sequence 4 were administered a single dose of 50 µg GSK2292767 in Period 1, 200 µg GSK2292767 in Period 2 and 1000 µg GSK2292767 in Period 3. The treatment was administered via ELLIPTA DPI. There was a period of 4 weeks between doses for an individual participant.
- Part A:Placebo/500 µg GSK2292767/2000 µg GSK2292767: Part A consisted of two cohorts each containing three treatment periods with four treatment sequences. Participants randomized to Sequence 5 were administered a single dose of placebo in Period 1, 500 µg GSK2292767 in Period 2 and 2000 µg GSK2292767 in Period 3. The treatment was administered via ELLIPTA DPI. There was a period of 4 weeks between doses for an individual participant.
- Part A:100 µg GSK2292767/Placebo/2000 µg GSK2292767: Part A consisted of two cohorts each containing three treatment periods with four treatment sequences. Participants randomized to Sequence 6 were administered a single dose of 100 ug GSK2292767 in Period 1, placebo in Period 2 and 2000 µg GSK2292767 in Period 3. The treatment was administered via ELLIPTA DPI. There was a period of 4 weeks between doses for an individual participant.
- Part A:100 µg GSK2292767/500 µg GSK2292767/Placebo: Part A consisted of two cohorts each containing three treatment periods with four treatment sequences. Participants randomized to Sequence 7 were administered a single dose of 100 µg GSK2292767 in Period 1, 500 µg GSK2292767 in Period 2 and placebo in Period 3. The treatment was administered via ELLIPTA DPI. There was a period of 4 weeks between doses for an individual participant.
- Part A:100 µg GSK2292767/500 µg GSK2292767/2000 µg GSK2292767: Part A consisted of two cohorts each containing three treatment periods with four treatment sequences. Participants randomized to Sequence 8 were administered a single dose of 100 µg GSK2292767 in Period 1, 500 µg GSK2292767 in Period 2 and 2000 µg GSK2292767 in Period 3. The treatment was administered via ELLIPTA DPI . There was a period of 4 weeks between doses for an individual participant.
- Part B:Placebo: Participants were administered once daily dose of placebo for 14 days via inhalation route using ELLIPTA DPI
- Part B:GSK2292767 2000 µg OD: Participants were administered 2000 µg GSK2292767 once daily for 14 days via inhalation route using ELLIPTA DPI
Period: Part A, Period (1 Day)
Arm/Group | Part A: Placebo/200 µg GSK2292767/1000 µg GSK2292767 | Part A:50 µg GSK2292767/Placebo/1000 µg GSK2292767 | Part A:50 µg GSK2292767/200 µg GSK2292767/Placebo | Part A:50 µg GSK2292767/200 µg GSK2292767/1000 µg GSK2292767 | Part A:Placebo/500 µg GSK2292767/2000 µg GSK2292767 | Part A:100 µg GSK2292767/Placebo/2000 µg GSK2292767 | Part A:100 µg GSK2292767/500 µg GSK2292767/Placebo | Part A:100 µg GSK2292767/500 µg GSK2292767/2000 µg GSK2292767 | Part B:Placebo | Part B:GSK2292767 2000 µg OD
Started | 7 | 4 | 5 | 5 | 4 | 4 | 4 | 4 | 0 | 0
Completed | 7 | 4 | 5 | 5 | 4 | 4 | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A,Washout Period 1(4 Weeks)
Arm/Group | Part A: Placebo/200 µg GSK2292767/1000 µg GSK2292767 | Part A:50 µg GSK2292767/Placebo/1000 µg GSK2292767 | Part A:50 µg GSK2292767/200 µg GSK2292767/Placebo | Part A:50 µg GSK2292767/200 µg GSK2292767/1000 µg GSK2292767 | Part A:Placebo/500 µg GSK2292767/2000 µg GSK2292767 | Part A:100 µg GSK2292767/Placebo/2000 µg GSK2292767 | Part A:100 µg GSK2292767/500 µg GSK2292767/Placebo | Part A:100 µg GSK2292767/500 µg GSK2292767/2000 µg GSK2292767 | Part B:Placebo | Part B:GSK2292767 2000 µg OD
Started | 7 | 4 | 5 | 5 | 4 | 4 | 4 | 4 | 0 | 0
Completed | 4 | 4 | 5 | 4 | 4 | 4 | 4 | 4 | 0 | 0
Not Completed | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A, Period 2 (1 Day)
Arm/Group | Part A: Placebo/200 µg GSK2292767/1000 µg GSK2292767 | Part A:50 µg GSK2292767/Placebo/1000 µg GSK2292767 | Part A:50 µg GSK2292767/200 µg GSK2292767/Placebo | Part A:50 µg GSK2292767/200 µg GSK2292767/1000 µg GSK2292767 | Part A:Placebo/500 µg GSK2292767/2000 µg GSK2292767 | Part A:100 µg GSK2292767/Placebo/2000 µg GSK2292767 | Part A:100 µg GSK2292767/500 µg GSK2292767/Placebo | Part A:100 µg GSK2292767/500 µg GSK2292767/2000 µg GSK2292767 | Part B:Placebo | Part B:GSK2292767 2000 µg OD
Started | 4 | 4 | 5 | 4 | 4 | 4 | 4 | 4 | 0 | 0
Completed | 3 | 4 | 5 | 4 | 4 | 4 | 4 | 4 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A,Washout Period 2 (4 Weeks)
Arm/Group | Part A: Placebo/200 µg GSK2292767/1000 µg GSK2292767 | Part A:50 µg GSK2292767/Placebo/1000 µg GSK2292767 | Part A:50 µg GSK2292767/200 µg GSK2292767/Placebo | Part A:50 µg GSK2292767/200 µg GSK2292767/1000 µg GSK2292767 | Part A:Placebo/500 µg GSK2292767/2000 µg GSK2292767 | Part A:100 µg GSK2292767/Placebo/2000 µg GSK2292767 | Part A:100 µg GSK2292767/500 µg GSK2292767/Placebo | Part A:100 µg GSK2292767/500 µg GSK2292767/2000 µg GSK2292767 | Part B:Placebo | Part B:GSK2292767 2000 µg OD
Started | 3 | 4 | 5 | 4 | 4 | 4 | 4 | 4 | 0 | 0
Completed | 3 | 4 | 4 | 2 | 4 | 4 | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A, Period 3 (1 Day)
Arm/Group | Part A: Placebo/200 µg GSK2292767/1000 µg GSK2292767 | Part A:50 µg GSK2292767/Placebo/1000 µg GSK2292767 | Part A:50 µg GSK2292767/200 µg GSK2292767/Placebo | Part A:50 µg GSK2292767/200 µg GSK2292767/1000 µg GSK2292767 | Part A:Placebo/500 µg GSK2292767/2000 µg GSK2292767 | Part A:100 µg GSK2292767/Placebo/2000 µg GSK2292767 | Part A:100 µg GSK2292767/500 µg GSK2292767/Placebo | Part A:100 µg GSK2292767/500 µg GSK2292767/2000 µg GSK2292767 | Part B:Placebo | Part B:GSK2292767 2000 µg OD
Started | 3 | 4 | 4 | 2 | 4 | 4 | 4 | 4 | 0 | 0
Completed | 3 | 4 | 4 | 2 | 4 | 4 | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (14 Days)
Arm/Group | Part A: Placebo/200 µg GSK2292767/1000 µg GSK2292767 | Part A:50 µg GSK2292767/Placebo/1000 µg GSK2292767 | Part A:50 µg GSK2292767/200 µg GSK2292767/Placebo | Part A:50 µg GSK2292767/200 µg GSK2292767/1000 µg GSK2292767 | Part A:Placebo/500 µg GSK2292767/2000 µg GSK2292767 | Part A:100 µg GSK2292767/Placebo/2000 µg GSK2292767 | Part A:100 µg GSK2292767/500 µg GSK2292767/Placebo | Part A:100 µg GSK2292767/500 µg GSK2292767/2000 µg GSK2292767 | Part B:Placebo | Part B:GSK2292767 2000 µg OD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data is presented for Part A and Part B. In Part B, 12 participants were included, 11 of them were taken from Part A and 1 additional participant only for Part B. Thus total number of participants included were 38 and not 49.
Groups:
- Part A:Placebo/200 µg GSK2292767/1000 µg GSK2292767: Part A consisted of two cohorts each containing three treatment periods with four treatment sequences. Participants randomized to Sequence 1 were administered a single dose of placebo in Period 1, 200 µg GSK2292767 in Period 2 and 1000 µg GSK2292767 in Period 3. The treatment was administered via ELLIPTA Dry Powder Inhaler (DPI). There was a period of 4 weeks between doses for an individual participant.
- Part B: Placebo: Participants were administered once daily dose of placebo for 14 days via inhalation route using ELLIPTA DPI
- Part B: GSK2292767 2000 µg OD: Participants were administered 2000 µg GSK2292767 once daily for 14 days via inhalation route using ELLIPTA DPI
- Total: Total of all reporting groups
Arm/Group | Part A:Placebo/200 µg GSK2292767/1000 µg GSK2292767 | Part A:50 µg GSK2292767/Placebo/1000 µg GSK2292767 | Part A:50 µg GSK2292767/200 µg GSK2292767/Placebo | Part A:50 µg GSK2292767/200 µg GSK2292767/1000 µg GSK2292767 | Part A:Placebo/500 µg GSK2292767/2000 µg GSK2292767 | Part A:100 µg GSK2292767/Placebo/2000 µg GSK2292767 | Part A:100 µg GSK2292767/500 µg GSK2292767/Placebo | Part A:100 µg GSK2292767/500 µg GSK2292767/2000 µg GSK2292767 | Part B: Placebo | Part B: GSK2292767 2000 µg OD | Total
Number analyzed (Participants) | 7 | 3 | 5 | 6 | 4 | 4 | 4 | 4 | 3 | 9 | 49
Age, Categorical [Count of Participants; unit: Participants] — All enrolled participants have been confirmed by site to have been at least 18 years at the time of screening. One participants has a derived age of 17 due to the way in which their partial birthdate was imputed.
  Participants
    <=18 years | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Between 18 and 65 years | 7 | 2 | 5 | 6 | 4 | 4 | 4 | 4 | 3 | 9 | 48
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 3 | 5 | 6 | 4 | 4 | 4 | 4 | 3 | 9 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian - Central/South Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 5 | 3 | 4 | 6 | 4 | 4 | 4 | 4 | 3 | 9 | 46

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Any Non-serious Adverse Event (nSAE) and Any Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinemia were categorized as SAE. Participants with 5 percent nSAEs and SAEs has been reported.
Time Frame: Up to 12 weeks
Population: Safety Population comprised of all randomized participants who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants administered a single dose of placebo using ELLIPTA DPI via inhalation route.
- 50 µg OD: Participants administered a single dose of 50 µg GSK2292767 via inhalation route using ELLIPTA DPI
- 100 µg OD: Participants administered a single dose of 100 µg GSK2292767 via inhalation route using ELLIPTA DPI
- 200 µg OD: Participants administered a single dose of 200 µg GSK2292767 via inhalation route using ELLIPTA DPI
- 500 µg OD: Participants administered a single dose of 500 µg GSK2292767 via inhalation route using ELLIPTA DPI
- 1000 µg OD: Participants administered a single dose of 1000 µg GSK2292767 via inhalation route using ELLIPTA DPI
- 2000 µg OD: Participants administered a single dose of 2000 µg GSK2292767 via inhalation route using ELLIPTA DPI
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 23 | 12 | 12 | 13 | 12 | 9 | 12
Participants
  nSAE | 6 | 9 | 6 | 7 | 6 | 4 | 5
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Number of Participants With Any AE and Any SAE
Description: as for outcome 1
Time Frame: Up to 4 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants were administered once daily dose of placebo for 14 days via inhalation route using ELLIPTA DPI
- 2000 µg OD: Participants were administered 2000 µg GSK2292767 once daily for 14 days via inhalation route using ELLIPTA DPI
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 3 | 9
Participants
  nSAE | 3 | 8
  SAE | 0 | 0

3. Primary Outcome: Part A: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure in part A was assessed in a semi supine position with a completely automated device. SBP and DBP measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment. Change from Baseline was defined as the value at indicated time point minus Baseline value.
Time Frame: Baseline, 30 minutes, 1, 6, 12 and 24 hours post-dose in each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 23 | 12 | 12 | 13 | 12 | 9 | 12
Millimeters of mercury
  DBP, 30 min | 0.3 (6.66) | 2.0 (6.48) | 2.4 (4.91) | 2.0 (5.23) | 2.5 (6.20) | -1.6 (5.36) | 1.9 (3.58)
  DBP, 1 hour | 0.8 (7.02) | 3.1 (4.98) | 3.8 (4.65) | 1.2 (3.63) | 4.1 (4.44) | -0.9 (7.72) | 0.8 (5.04)
  DBP, 6 hour | 0.1 (5.48) | 0.3 (7.41) | 1.8 (3.84) | 1.9 (7.04) | 3.2 (6.22) | -2.0 (2.83) | 3.1 (7.93)
  DBP, 12 hour | 2.3 (6.36) | 3.1 (6.72) | 2.9 (3.45) | 4.0 (7.92) | 2.3 (6.41) | 0.7 (4.39) | 3.1 (7.76)
  DBP, 24 hour | -1.3 (6.81) | 0.6 (6.32) | 1.5 (3.90) | 3.6 (8.03) | 3.6 (4.21) | -2.9 (5.62) | -0.1 (5.12)
  SBP, 30 min | -3.2 (6.28) | -0.2 (5.06) | -3.9 (9.67) | 0.8 (5.16) | -2.3 (6.20) | -6.1 (4.73) | -3.3 (5.85)
  SBP, 1 hour | -3.4 (7.72) | -1.5 (4.74) | -5.6 (8.07) | -3.4 (7.01) | -2.2 (6.53) | -7.1 (9.06) | -3.9 (8.38)
  SBP, 6 hour | 1.3 (8.79) | 0.7 (8.23) | -3.8 (9.03) | 4.5 (7.92) | 2.8 (6.34) | -0.3 (7.48) | -0.8 (5.86)
  SBP, 12 hour | 3.9 (6.65) | 3.3 (6.52) | -1.3 (8.65) | 3.6 (4.93) | 5.0 (9.53) | 1.6 (4.03) | 3.3 (7.33)
  SBP, 24 hour | -0.7 (6.19) | -0.9 (7.54) | -5.3 (5.26) | 0.0 (8.67) | -1.5 (6.78) | -4.3 (5.74) | -2.8 (5.77)

4. Primary Outcome: Part B: Change From Baseline in SBP and DBP
Description: Blood pressure in part B were assessed in semi supine position with a completely automated device. SBP and DBP preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as measurements done on Day -1. Change from Baseline was defined as the value at indicated time point minus Baseline value.
Time Frame: Baseline, Pre-dose on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14, 24 hours post-dose on Day 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 3 | 9
Millimeters of mercury
  DBP, Day 2, pre-dose | -6.0 (10.15) | -3.0 (4.72)
  DBP, Day 3, pre-dose | -8.3 (9.45) | -1.3 (5.85)
  DBP, Day 4, pre-dose | -7.3 (12.10) | -3.4 (4.90)
  DBP, Day 5, pre-dose | -10.7 (11.72) | -2.2 (5.09)
  DBP, Day 6, pre-dose | -7.7 (10.02) | -3.7 (4.72)
  DBP, Day 7, pre-dose | -8.3 (9.45) | -2.3 (3.57)
  DBP, Day 8, pre-dose | -5.7 (12.42) | -4.3 (3.91)
  DBP, Day 9, pre-dose | -6.3 (11.93) | -2.8 (4.02)
  DBP, Day 10, pre-dose | -8.7 (11.93) | -0.6 (6.21)
  DBP, Day 11, pre-dose | -9.3 (12.74) | -2.1 (4.46)
  DBP, Day 12, pre-dose | -7.3 (7.51) | -2.9 (4.23)
  DBP, Day 13, pre-dose | -7.0 (10.58) | -3.0 (5.43)
  DBP, Day 14, pre-dose | -8.3 (10.97) | -3.2 (3.83)
  DBP, Day 14, 24 hours | -1.3 (1.53) | -1.0 (5.17)
  SBP, Day 2, pre-dose | 3.3 (11.24) | -5.4 (7.60)
  SBP, Day 3, pre-dose | -0.7 (9.07) | -0.1 (8.70)
  SBP, Day 4, pre-dose | 2.3 (10.50) | -4.1 (7.75)
  SBP, Day 5, pre-dose | -1.0 (9.85) | -5.1 (8.74)
  SBP, Day 6, pre-dose | -1.7 (8.50) | -7.2 (7.26)
  SBP, Day 7, pre-dose | -4.7 (5.86) | -5.0 (9.50)
  SBP, Day 8, pre-dose | -1.3 (8.08) | -7.6 (10.01)
  SBP, Day 9, pre-dose | 0.0 (3.61) | -5.8 (4.27)
  SBP, Day 10, pre-dose | -4.7 (5.13) | -5.2 (6.65)
  SBP, Day 11, pre-dose | -6.3 (5.51) | -4.4 (9.06)
  SBP, Day 12, pre-dose | -6.3 (4.73) | -5.4 (6.54)
  SBP, Day 13, pre-dose | 2.3 (4.93) | -4.9 (6.51)
  SBP, Day 14, pre-dose | -1.7 (7.57) | -4.6 (7.33)
  SBP, Day 14, 24 hours | -0.7 (2.08) | -3.7 (6.71)

5. Primary Outcome: Part A: Change From Baseline in Heart Rate
Description: Heart rate in part A was assessed in a semi supine position with a completely automated device. Heart rate measurement was preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as latest pre-dose measurement. Change from Baseline was defined as the value at indicated time point minus Baseline value.
Time Frame: Baseline, 30 minutes, 1, 6, 12 and 24 hours post-dose in each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 23 | 12 | 12 | 13 | 12 | 9 | 12
Beats per minute
  30 min | -5.3 (5.39) | -5.8 (5.40) | -8.9 (8.46) | -6.1 (5.25) | -6.3 (5.37) | -12.4 (6.80) | -6.1 (7.24)
  1 hour | -8.0 (5.60) | -4.8 (3.57) | -9.0 (8.90) | -7.2 (5.27) | -4.3 (7.63) | -13.0 (7.98) | -9.8 (7.55)
  6 hour | 4.3 (9.45) | 4.3 (5.58) | 1.0 (9.55) | 4.9 (5.42) | 7.4 (6.37) | -1.3 (7.42) | 2.4 (7.98)
  12 hour | 4.2 (7.11) | 6.4 (7.80) | -0.3 (10.17) | 3.7 (6.24) | 3.7 (5.85) | -1.8 (8.61) | 5.3 (10.38)
  24 hour | -2.3 (6.24) | -1.7 (6.69) | -1.8 (8.70) | -3.0 (7.23) | -1.8 (8.02) | -6.9 (5.88) | -4.0 (8.18)

6. Primary Outcome: Part B: Change From Baseline in Heart Rate
Description: Heart rate in part B was assessed in a semi supine position with a completely automated device. Heart rate measurement was preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as latest pre-dose measurement. Change from Baseline was defined as the value at indicated time point minus Baseline value.
Time Frame: Baseline, Pre-dose on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14, 24 hours post-dose on Day 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 3 | 9
Beats per minute
  Day 2, pre-dose | -0.3 (6.11) | -0.7 (7.14)
  Day 3, pre-dose | 3.0 (6.56) | 0.0 (6.76)
  Day 4, pre-dose | 6.7 (11.50) | -2.2 (8.03)
  Day 5, pre-dose | -2.3 (9.45) | -3.2 (9.26)
  Day 6, pre-dose | -2.7 (8.14) | -6.4 (7.80)
  Day 7, pre-dose | 3.7 (9.07) | -0.8 (11.12)
  Day 8, pre-dose | 4.7 (13.50) | -3.2 (5.85)
  Day 9, pre-dose | 1.7 (5.13) | -3.4 (8.49)
  Day 10, pre-dose | 1.0 (11.79) | -2.7 (10.28)
  Day 11, pre-dose | -1.3 (14.64) | -2.8 (11.98)
  Day 12, pre-dose | -5.7 (7.23) | -4.9 (6.47)
  Day 13, pre-dose | 4.0 (15.00) | -4.4 (6.13)
  Day 14, pre-dose | 6.0 (11.27) | -5.8 (9.36)
  Day 14, 24 hours | -2.3 (7.57) | -2.2 (7.56)

7. Primary Outcome: Part A: Change From Baseline in Respiratory Rate
Description: Respiratory rate in part A was assessed in a semi supine position after 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as measurements done on Day -1. Change from Baseline was defined as the value at indicated time point minus Baseline value. Baseline was defined as latest pre-dose measurement. Change from Baseline was defined as the value at indicated time point minus Baseline value.
Time Frame: Baseline, 30 minutes, 1, 6, 12 and 24 hours post-dose in each treatment period
Population: Safety Population
Measure: Median (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 23 | 12 | 12 | 13 | 12 | 9 | 12
Breaths per minute
  30 min | -0.2 (1.78) | -1.1 (2.81) | -1.5 (1.98) | 0.8 (2.48) | 0.3 (2.01) | 0.3 (2.74) | -0.2 (1.95)
  1 hour | -0.3 (2.27) | -1.0 (2.76) | -1.2 (2.17) | 0.8 (2.03) | 0.6 (2.23) | -0.3 (2.35) | -0.8 (2.41)
  6 hour | 0.1 (2.18) | 0.0 (3.67) | 1.0 (1.95) | 1.0 (2.97) | 0.8 (3.33) | 0.6 (2.74) | 0.3 (2.23)
  12 hour | 0.7 (2.31) | 0.7 (3.11) | -0.4 (2.43) | 1.3 (2.14) | 0.6 (2.75) | 0.3 (2.55) | -0.3 (1.86)
  24 hour | -0.6 (2.29) | -0.9 (3.20) | -1.0 (2.63) | 0.4 (2.50) | -0.8 (2.08) | -0.8 (3.15) | -0.4 (1.68)

8. Primary Outcome: Part B: Change From Baseline in Respiratory Rate
Description: Respiratory rate in part B was assessed in a semi supine position after 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as measurements done on Day -1. Change from Baseline was defined as the value at indicated time point minus Baseline value. Baseline was defined as latest pre-dose measurement. Change from Baseline was defined as the value at indicated time point minus Baseline value.
Time Frame: Baseline, Pre-dose on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14, 24 hours post-dose on Day 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 3 | 9
Breaths per minute
  Day 2, pre-dose | -2.3 (0.58) | -0.6 (3.17)
  Day 3, pre-dose | -2.3 (2.31) | -1.0 (3.20)
  Day 4, pre-dose | -2.3 (2.08) | -0.3 (2.96)
  Day 5, pre-dose | -2.7 (2.31) | -1.4 (2.65)
  Day 6, pre-dose | -2.7 (0.58) | -1.6 (2.92)
  Day 7, pre-dose | -2.3 (2.31) | -0.8 (2.59)
  Day 8, pre-dose | -2.7 (0.58) | -0.7 (2.45)
  Day 9, pre-dose | -2.0 (2.00) | 0.1 (2.98)
  Day 10, pre-dose | -1.7 (2.31) | -1.2 (2.54)
  Day 11, pre-dose | -3.3 (0.58) | -0.9 (3.62)
  Day 12, pre-dose | -2.3 (1.15) | -1.0 (2.74)
  Day 13, pre-dose | -1.3 (1.15) | -0.1 (3.06)
  Day 14, pre-dose | -2.0 (1.73) | -1.1 (2.89)
  Day 14, 24 hours | -2.3 (1.53) | -1.1 (2.26)

9. Primary Outcome: Part A: Change From Baseline in Tympanic Temperature
Description: Tympanic temperature in part A was assessed in semi supine position after 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as measurements done on Day -1. Change from Baseline was defined as the value at indicated time point minus Baseline value. Baseline was defined as latest pre-dose measurement. Change from Baseline was defined as the value at indicated time point minus Baseline value.
Time Frame: Baseline, 30 minutes, 1, 6, 12 and 24 hours post-dose in each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 23 | 12 | 12 | 13 | 12 | 9 | 12
Celsius
  30 min | 0.03 (0.313) | 0.07 (0.210) | 0.04 (0.574) | 0.05 (0.395) | -0.05 (0.366) | 0.03 (0.287) | 0.16 (0.385)
  1 hour | -0.10 (0.348) | 0.06 (0.173) | 0.05 (0.498) | -0.06 (0.287) | 0.05 (0.478) | 0.12 (0.311) | 0.10 (0.449)
  6 hour | 0.20 (0.390) | 0.08 (0.259) | 0.18 (0.566) | 0.07 (0.446) | 0.17 (0.409) | 0.14 (0.361) | 0.19 (0.493)
  12 hour | 0.14 (0.478) | 0.31 (0.370) | 0.27 (0.542) | 0.26 (0.355) | 0.20 (0.591) | 0.46 (0.400) | 0.18 (0.622)
  24 hour | -0.06 (0.375) | -0.02 (0.233) | -0.02 (0.513) | 0.03 (0.287) | 0.07 (0.392) | 0.11 (0.326) | 0.02 (0.497)

10. Primary Outcome: Part B: Change From Baseline in Tympanic Temperature
Description: Tympanic temperature in part B was assessed in semi supine position after 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as measurements done on Day -1. Change from Baseline was defined as the value at indicated time point minus Baseline value. Baseline was defined as latest pre-dose measurement. Change from Baseline was defined as the value at indicated time point minus Baseline value.
Time Frame: Baseline, Pre-dose on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14, 24 hours post-dose on Day 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 3 | 9
Celsius
  Day 2, pre-dose | 0.17 (0.058) | 0.26 (0.477)
  Day 3, pre-dose | 0.03 (0.379) | 0.37 (0.450)
  Day 4, pre-dose | 0.13 (0.153) | 0.26 (0.416)
  Day 5, pre-dose | 0.13 (0.404) | 0.34 (0.445)
  Day 6, pre-dose | 0.10 (0.265) | 0.31 (0.322)
  Day 7, pre-dose | -0.10 (0.100) | 0.41 (0.448)
  Day 8, pre-dose | -0.27 (0.231) | 0.29 (0.462)
  Day 9, pre-dose | -0.03 (0.153) | 0.21 (0.326)
  Day 10, pre-dose | 0.13 (0.451) | 0.31 (0.392)
  Day 11, pre-dose | 0.13 (0.306) | 0.34 (0.343)
  Day 12, pre-dose | 0.00 (0.265) | 0.32 (0.415)
  Day 13, pre-dose | 0.07 (0.513) | 0.33 (0.466)
  Day 14, pre-dose | 0.17 (0.115) | 0.32 (0.458)
  Day 14, 24 hours | 0.17 (0.115) | 0.32 (0.502)

11. Primary Outcome: Part A: Maximal Amount of Air Forcefully Exhaled in 1 Second (FEV1)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured using spirometry at the indicated time. FEV1 measurements were repeated until three technically acceptable measurements (within 150 milliliter [mL] of each other) were made. Data for FEV1 for part A is presented here.
Time Frame: Day 1 (pre-dose and 1 hour)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 23 | 12 | 12 | 13 | 12 | 9 | 12
Liters
  Pre-dose | 4.389 (0.6781) | 4.044 (0.6717) | 4.768 (0.8348) | 3.896 (0.7292) | 4.288 (0.5288) | 4.036 (0.4806) | 4.391 (0.5072)
  1 hour | 4.347 (0.6781) | 4.028 (0.7177) | 4.461 (0.4693) | 3.811 (0.6757) | 4.223 (0.5153) | 4.024 (0.5971) | 4.435 (0.5851)

12. Primary Outcome: Part B: Maximal Amount of Air Forcefully Exhaled in 1 Second (FEV1)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured using spirometry at the indicated time. Existing spirometry equipment was used. FEV1 measurements were repeated until three technically acceptable measurements (within 150 mL of each other) were made. Data for FEV1 for part B is presented here.
Time Frame: Up to Day 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 3 | 9
Liters
  Day -1 | 4.333 (0.1739) | 4.570 (0.6275)
  Day 1,pre-dose | 4.277 (0.0987) | 4.408 (0.6852)
  Day 1,1 hour | 4.323 (0.0981) | 4.413 (0.6931)
  Day 2,pre-dose | 4.357 (0.0551) | 4.446 (0.7230)
  Day 2,1 hour | 4.373 (0.0569) | 4.486 (0.6828)
  Day 3,pre-dose | 4.407 (0.1504) | 4.474 (0.6999)
  Day 3,1 hour | 4.460 (0.2771) | 4.493 (0.6548)
  Day 4,pre-dose | 4.447 (0.1159) | 4.483 (0.7241)
  Day 4,1 hour | 4.307 (0.1060) | 4.519 (0.7444)
  Day 5,pre-dose | 4.290 (0.1082) | 4.494 (0.8042)
  Day 5,1 hour | 4.480 (0.2600) | 4.486 (0.7647)
  Day 6,pre-dose | 4.300 (0.0173) | 4.498 (0.7086)
  Day 6,1 hour | 4.533 (0.3177) | 4.573 (0.7994)
  Day 7,pre-dose | 4.467 (0.2386) | 4.503 (0.8559)
  Day 7,1 hour | 4.400 (0.2207) | 4.581 (0.8018)
  Day 8,pre-dose | 4.383 (0.0351) | 4.449 (0.7952)
  Day 8,1 hour | 4.440 (0.1229) | 4.572 (0.6952)
  Day 9,pre-dose | 4.483 (0.2458) | 4.512 (0.7483)
  Day 9,1 hour | 4.470 (0.1179) | 4.627 (0.7737)
  Day 10,pre-dose | 4.443 (0.1419) | 4.473 (0.6942)
  Day 10,1 hour | 4.583 (0.1914) | 4.582 (0.7609)
  Day 11,pre-dose | 4.423 (0.1422) | 4.570 (0.7944)
  Day 11,1 hour | 4.463 (0.2540) | 4.609 (0.7460)
  Day 12,pre-dose | 4.417 (0.1258) | 4.599 (0.7469)
  Day 12,1 hour | 4.440 (0.0917) | 4.600 (0.7029)
  Day 13,pre-dose | 4.400 (0.2252) | 4.514 (0.7352)
  Day 13,1 hour | 4.653 (0.2146) | 4.768 (0.7609)
  Day 14,pre-dose | 4.533 (0.0666) | 4.541 (0.8512)
  Day 14,1 hour | 4.557 (0.1701) | 4.609 (0.8102)

13. Primary Outcome: Part A: Forced Vital Capacity (FVC)
Description: FVC is a measure of lung function and is defined as total amount of air that can be exhaled during FEV1 test. FVC was planned to measured using spirometry. The FVC need to be normal at screening and is part of the Forced Expiratory ratio (FEV1/FVC) which should lie between 0.7-0.8 to indicate no chronic obstruction or restriction. The FVC was therefore only used at screening and requires no ongoing analysis during the study. All other indications of obstruction in the study, e.g. paradoxical bronchospasm was provided by the FEV1. The FVC therefore require no analysis.
Time Frame: Day 1 (pre-dose and 1 hour)
Population: Safety Population. Data was not collected for this outcome as FVC was used only at screening and no further analysis during the study was required.
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Part B: Forced Vital Capacity (FVC)
Description: as for outcome 13
Time Frame: Day 1 (pre-dose and 1 hour)
Population: as for outcome 13
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Part A: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Triplicate/Single 12-lead ECG was obtained using an automated ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTFc intervals. Number of participants with abnormal clinically significant and abnormal-not clinically significant values at any time post-Baseline is presented.
Time Frame: Day 1 of each treatment period
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 23 | 12 | 12 | 13 | 12 | 9 | 12
Participants
  Abnormal - not clinically significant | 2 | 2 | 1 | 0 | 1 | 0 | 1
  Abnormal - clinically significant | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Part B: Number of Participants With ECG Abnormalities
Description: as for outcome 15
Time Frame: Pre-dose on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14, 24 hours post-dose on Day 14
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 3 | 9
Participants
  Abnormal - not clinically significant | 1 | 2
  Abnormal - clinically significant | 0 | 0

17. Primary Outcome: Part A: Number of Participants With Clinical Chemistry Values of Potential Clinical Importance Criteria (PCC)
Description: Number of participants with clinical chemistry values that changed from normal to high or low in part A are presented. Chemistry parameters for which PCC values were identified were: Alkaline Phosphatase, Alanine Amino Transferase, aspartate aminotransferase, Total Bilirubin, calcium, glucose, potassium and Sodium.
Time Frame: 24 hours post-dose in each treatment period.
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 23 | 12 | 12 | 13 | 12 | 9 | 12
Participants
  Alkaline Phosphatase; to high | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Amino Transferase; to high | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Aspartate Amino Transferase; to high | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin; to high | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; to high | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; to low | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; to high | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Glucose; to low | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium; to high | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium; to low | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium; to high | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium; to low | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Part B: Number of Participants With Clinical Chemistry Values of PCC
Description: Number of participants with clinical chemistry values that changed from normal to high or low in part B are presented. Chemistry parameters for which PCC values were identified were: Alkaline Phosphatase, Alanine Amino Transferase, aspartate aminotransferase, Total Bilirubin, calcium, glucose, potassium and Sodium. Only participants with data available at specified time points were analyzed (represented by n=X in category titles)
Time Frame: Pre-dose on Days 2, 4, 6, 8, 10, 12, and 14, 24 hours post-dose on Day 14
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 3 | 9
Participants
  Alkaline Phosphatase,Day 2;to high,n=3,9 | 0 | 0
  Alkaline Phosphatase,Day 4;to high,n=3,9 | 0 | 0
  Alkaline Phosphatase,Day 6;to high,n=3,9 | 0 | 0
  Alkaline Phosphatase,Day 8;to high,n=3,9 | 0 | 0
  Alkaline Phosphatase,Day 10;to high,n=3,9 | 0 | 0
  Alkaline Phosphatase,Day 12;to high,n=3,9 | 0 | 0
  Alkaline Phosphatase,Day 14,pre-dose;to high,n=3,9 | 0 | 0
  Alkaline Phosphatase,Day 14,24 hour;to high,n=3,9 | 0 | 0
  Alanine Amino Transferase,Day 2;to high,n=3,9 | 0 | 0
  Alanine Amino Transferase,Day 4;to high,n=3,9 | 0 | 0
  Alanine Amino Transferase,Day 6;to high,n=3,9 | 0 | 0
  Alanine Amino Transferase,Day 8;to high,n=3,9 | 0 | 0
  Alanine Amino Transferase,Day 10;to high,n=3,9 | 0 | 0
  Alanine Amino Transferase,Day 12;to high,n=3,9 | 0 | 0
  Alanine Amino Transferase,Day 14,pre dose;to n=3,9 | 0 | 0
  Alanine Amino Transferase,Day 14,24 hour;to hn=3,9 | 0 | 0
  Aspartate Amino Transferase,Day 2;to high,n=3,8: number analyzed (Participants) | 3 | 8
  Aspartate Amino Transferase,Day 2;to high,n=3,8 | 0 | 0
  Aspartate Amino Transferase,Day 4;to high,n=3,9 | 0 | 0
  Aspartate Amino Transferase,Day 6;to high,n=3,9 | 0 | 0
  Aspartate Amino Transferase,Day 8;to high,n=3,9 | 0 | 0
  Aspartate Amino Transferase,Day 10;to high,n=3,9 | 0 | 0
  Aspartate Amino Transferase,Day 12;to high,n=3,9 | 0 | 0
  Aspartate Amino Transferase,Day 14,pre dose;n=2,9: number analyzed (Participants) | 2 | 9
  Aspartate Amino Transferase,Day 14,pre dose;n=2,9 | 0 | 0
  Aspartate Amino Transferase,Day 14,24 hour,n=3,8: number analyzed (Participants) | 3 | 8
  Aspartate Amino Transferase,Day 14,24 hour,n=3,8 | 0 | 0
  Total Bilirubin,Day 2,;to high,n=3,9 | 0 | 0
  Total Bilirubin,Day 4;to high,n=3,9 | 0 | 0
  Total Bilirubin,Day 6;to high,n=3,9 | 0 | 0
  Total Bilirubin,Day 8;to high,n=3,9 | 0 | 0
  Total Bilirubin,Day 10;to high,n=3,9 | 0 | 0
  Total Bilirubin,Day 12;to high,n=3,9 | 0 | 0
  Total Bilirubin,Day 14,pre dose,n=3,9 | 0 | 0
  Total Bilirubin,Day 14,24 hours,n=3,9 | 0 | 0
  Calcium,Day 2;to high,n=3,9 | 0 | 0
  Calcium,Day 2;to low,n=3,9 | 0 | 0
  Calcium,Day 4;to high,n=3,9 | 0 | 0
  Calcium,Day 4;to low,n=3,9 | 0 | 0
  Calcium,Day 6;to high,n=3,9 | 0 | 0
  Calcium,Day 6;to low,n=3,9 | 0 | 0
  Calcium,Day 8;to high,n=3,9 | 0 | 0
  Calcium,Day 8;to low,n=3,9 | 0 | 0
  Calcium,Day 10;to high,n=3,9 | 0 | 0
  Calcium,Day 10;to low,n=3,9 | 0 | 0
  Calcium,Day 12;to high,n=3,9 | 0 | 0
  Calcium,Day 12;to low,n=3,9 | 0 | 0
  Calcium,Day 14,pre dose,to high,n=3,9 | 0 | 0
  Calcium,Day 14,pre dose,to low,n=3,9 | 0 | 0
  Calcium,Day 14,24 hour,to high,n=3,9 | 0 | 0
  Calcium,Day 14,24 hour,to low,n=3,9 | 0 | 0
  Glucose,Day 2;to high,n=3,9 | 0 | 0
  Glucose,Day 2;to low,n=3,9 | 0 | 0
  Glucose,Day 4;to high,n=3,9 | 0 | 0
  Glucose,Day 4;to low,n=3,9 | 0 | 0
  Glucose,Day 6;to high,n=3,9 | 0 | 0
  Glucose,Day 6;to low, n=3,9 | 0 | 0
  Glucose,Day 8;to high,n=3,9 | 0 | 0
  Glucose,Day 8;to low,n=3,9 | 0 | 0
  Glucose,Day 10;to high,n=3,9 | 0 | 0
  Glucose,Day 10;to low,,n=3,9 | 0 | 0
  Glucose,Day 12;to high,n=3,9 | 0 | 0
  Glucose,Day 12;to low,n=3,9 | 0 | 0
  Glucose,Day 14;pre dose,to high,n=3,9 | 0 | 0
  Glucose,Day 14;pre dose,to low,n=3,9 | 0 | 0
  Glucose,Day 14;24 hours,to high,n=3,9 | 0 | 0
  Glucose,Day 14;24 hours,to low,n=3,9 | 0 | 0
  Potassium,Day 2;to high,n=3,9 | 0 | 0
  Potassium,Day 2;to low,n=3,9 | 0 | 0
  Potassium,Day 4;to high,n=3,9 | 0 | 0
  Potassium,Day 4,n=3,9 | 0 | 0
  Potassium,Day 6;to high,n=3,9 | 0 | 0
  Potassium,Day 6,to low,n=3,9 | 0 | 0
  Potassium,Day 8;to high,n=3,9 | 0 | 0
  Potassium,Day 8, to low,n=3,9 | 0 | 0
  Potassium,Day 10;to high,,n=3,9 | 0 | 0
  Potassium,Day 10,to low,n=3,9 | 0 | 0
  Potassium,Day 12;to high,,n=3,9 | 0 | 0
  Potassium,Day 12,to low,n=3,9 | 0 | 0
  Potassium,Day 14,pre dose,to high,n=3,9 | 0 | 0
  Potassium,Day 14,pre dose,to low,n=3,9 | 0 | 0
  Potassium,Day 14,24 hour ,to low,n=3,9 | 0 | 0
  Potassium,Day 14,24 hour,to low,n=3,9 | 0 | 0
  Sodium,Day 2, to high,n=3,9 | 0 | 0
  Sodium,Day 2, to low,n=3,9 | 0 | 0
  Sodium,Day 4, to high,n=3,9 | 0 | 0
  Sodium,Day 4, to low,n=3,9 | 0 | 0
  Sodium,Day 6, to high,n=3,9 | 0 | 0
  Sodium,Day 6, to low,n=3,9 | 0 | 0
  Sodium,Day 8, to high,n=3,9 | 0 | 0
  Sodium,Day 8, to low,n=3,9 | 0 | 0
  Sodium,Day 10, to high,n=3,9 | 0 | 0
  Sodium,Day 10, to low,n=3,9 | 0 | 0
  Sodium,Day 12, to high,n=3,9 | 0 | 0
  Sodium,Day 12, to low,n=3,9 | 0 | 0
  Sodium,Day 14,pre dose, to high,n=3,9 | 0 | 0
  Sodium,Day 14,pre dose, to low,n=3,9 | 0 | 0
  Sodium,Day 14,24 hour, to high,n=3,9 | 0 | 0
  Sodium,Day 14,24 hour, to low,n=3,9 | 0 | 0

19. Primary Outcome: Part A: Number of Participants With Hematology Values of PCC
Description: Number of participants with hematology parameters of PCC which shifted from normal to high in part A are presented. Hematology parameters for which PCC values were identified were: Hemoglobin, Hematocrit, Lymphocytes, Total Neutrophils, Platelet count and White Blood Cell (WBC) Count. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles)
Time Frame: 24 hours post-dose in each treatment period
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 23 | 12 | 12 | 13 | 12 | 9 | 12
Participants
  Hemoglobin; to high,n=23,12,12,13,12,9,12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit; to high,n=23,12,12,13,12,9,12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes; to low,n=23,12,12,13,12,9,12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Neutrophils; to low,n=23,12,12,13,12,9,12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count;to high;n=23, 12, 11, 13, 11, 9, 11: number analyzed (Participants) | 23 | 12 | 11 | 13 | 11 | 9 | 11
  Platelet count;to high;n=23, 12, 11, 13, 11, 9, 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count; to low;n=23, 12, 11, 13, 11, 9, 11: number analyzed (Participants) | 23 | 12 | 11 | 13 | 11 | 9 | 11
  Platelet count; to low;n=23, 12, 11, 13, 11, 9, 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC count,to high,n=23, 12, 12, 13, 12, 9, 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC count,to low,n=23, 12, 12, 13, 12, 9, 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Primary Outcome: Part B: Number of Participants With Hematology Values of PCC
Description: Number of participants with hematology parameters of PCC which shifted from normal to high in part B are presented. Hematology parameters for which PCC values were identified were: Hemoglobin, Hematocrit, Lymphocytes, Total Neutrophils, Platelet count and WBC count
Time Frame: Pre-dose on Days 2, 4, 6, 8, 10, 12, and 14, 24 hours post-dose on Day 14
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2000 µg OD
Number analyzed (Participants) | 3 | 9
Participants
  Hemoglobin,Day 2 | 0 | 0
  Hemoglobin,Day 4 | 0 | 0
  Hemoglobin,Day 6 | 0 | 0
  Hemoglobin,Day 8 | 0 | 0
  Hemoglobin,Day 10 | 0 | 0
  Hemoglobin,Day 12 | 0 | 0
  Hemoglobin,Day 14,pre dose | 0 | 0
  Hemoglobin,Day 14,24 hour | 0 | 0
  Hematocrit,Day 2 | 0 | 0
  Hematocrit,Day 4 | 0 | 0
  Hematocrit,Day 6 | 0 | 0
  Hematocrit,Day 8 | 0 | 0
  Hematocrit,Day 10 | 0 | 0
  Hematocrit,Day 12 | 0 | 0
  Hematocrit,Day 14,pre dose | 0 | 0
  Hematocrit,Day 14,24 hour | 0 | 0
  Lymphocytes,Day 2 | 0 | 0
  Lymphocytes,Day 4 | 0 | 0
  Lymphocytes,Day 6 | 0 | 0
  Lymphocytes,Day 8 | 0 | 0
  Lymphocytes,Day 10 | 0 | 0
  Lymphocytes,Day 12 | 0 | 0
  Lymphocytes,Day 14,pre dose | 0 | 0
  Lymphocytes,Day 14,24 hour | 0 | 0
  Total Neutrophils,Day 2 | 0 | 0
  Total Neutrophils,Day 4 | 0 | 0
  Total Neutrophils,Day 6 | 0 | 0
  Total Neutrophils,Day 8 | 0 | 0
  Total Neutrophils,Day 10 | 0 | 0
  Total Neutrophils,Day 12 | 0 | 0
  Total Neutrophils,Day 14,pre dose | 0 | 0
  Total Neutrophils,Day 14,24 hour | 0 | 0
  Platelet count,Day 2 | 0 | 0
  Platelet count,Day 4 | 0 | 0
  Platelet count,Day 6 | 0 | 0
  Platelet count,Day 8 | 0 | 0
  Platelet count,Day 10 | 0 | 0
  Platelet count,Day 12 | 0 | 0
  Platelet count,Day 14,pre dose | 0 | 0
  Platelet count,Day 14,24 hour | 0 | 0
  WBC count,Day 2 | 0 | 0
  WBC count,Day 4 | 0 | 0
  WBC count,Day 6 | 0 | 0
  WBC count,Day 8 | 0 | 0
  WBC count,Day 10 | 0 | 0
  WBC count,Day 12 | 0 | 0
  WBC count,Day 14,pre dose | 0 | 0
  WBC count,Day 14,24 hour | 0 | 0

21. Secondary Outcome: Part A: Area Under the Plasma Drug Concentration Versus Time Curve (AUC) From Zero to Time t (AUC [0 to t]), AUC From Zero to 24 Hours (AUC [0 to 24]) and AUC From Zero to Infinity (AUC [0 to Inf]) of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Data for AUC (0 to t), AUC (0 to 24) and AUC (0 to inf) of GSK2292767 for part A is presented. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). Pharmacokinetic population comprised of participants in the 'All participant' population for whom a pharmacokinetic sample was obtained and analyzed.
Time Frame: Pre-dose (5 minutes (min), 30 min, 45 min, 1 hour (hr), 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr post dose in each of the 3 treatment periods
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picograms per milliliter
Arm/Group | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 12 | 12 | 13 | 12 | 9 | 12
Hours*picograms per milliliter
  AUC (0-24);n=0,2,5,10,8,11: number analyzed (Participants) | 0 | 2 | 5 | 10 | 8 | 11
  AUC (0-24);n=0,2,5,10,8,11 |  | 596.1161 (10.0) | 721.9301 (57.9) | 2460.3695 (70.3) | 3689.7545 (36.0) | 7781.2593 (52.5)
  AUC(0-inf);n=0,2,5,7,6,10: number analyzed (Participants) | 0 | 2 | 5 | 7 | 6 | 10
  AUC(0-inf);n=0,2,5,7,6,10 |  | 596.4042 (10.1) | 724.6058 (57.8) | 2211.9120 (81.5) | 3709.6509 (40.6) | 8383.6427 (57.8)
  AUC (0-t);n=12,12,12,12,9,12: number analyzed (Participants) | 12 | 12 | 12 | 12 | 9 | 12
  AUC (0-t);n=12,12,12,12,9,12 | 69.5822 (133.1) | 337.0775 (48.3) | 633.3267 (59.6) | 2164.3817 (72.3) | 3440.6354 (37.1) | 7758.9831 (50.9)
Statistical Analysis 1: Comparison: 50 µg OD vs 100 µg OD; Test type: Other; Ratio = 0.41, 90% CI 2-sided [0.27 to 0.61], Standard Error of Mean 0.243 — AUC(0-t). Standard error of mean was on logged scale
Statistical Analysis 2: Comparison: 100 µg OD vs 200 µg OD; Test type: Other; Ratio = 0.98, 90% CI 2-sided [0.65 to 1.47], Standard Error of Mean 0.243 — AUC(0-t).Standard error of mean was on logged scale
Statistical Analysis 3: Comparison: 100 µg OD vs 500 µg OD; Test type: Other; Ratio = 1.33, 90% CI 2-sided [1.01 to 1.74], Standard Error of Mean 0.161 — AUC(0-t).Standard error of mean was on logged scale
Statistical Analysis 4: Comparison: 100 µg OD vs 1000 µg OD; Test type: Other; Ratio = 1.06, 90% CI 2-sided [0.69 to 1.62], Standard Error of Mean 0.255 — AUC(0-t).Standard error of mean was on logged scale
Statistical Analysis 5: Comparison: 100 µg OD vs 2000 µg OD; Test type: Other; Ratio = 1.25, 90% CI 2-sided [0.95 to 1.64], Standard Error of Mean 0.161 — AUC(0-t).Standard error of mean was on logged scale

22. Secondary Outcome: Part B: AUC (0 to t), AUC (0 to 24) and AUC (0 to Inf) of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Data for AUC (0 to t), AUC (0 to 24) and AUC (0 to inf) of GSK2292767 for part B is presented. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Pre-dose, 5 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 8 and 12hours post dose on Day 1; pre-dose, 5 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 8 and 12hours post dose on Day 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picograms per milliliter
Arm/Group | 2000 µg OD
Number analyzed (Participants) | 9
Hours*picograms per milliliter
  AUC (0-24); Day 1; n=8: number analyzed (Participants) | 8
  AUC (0-24); Day 1; n=8 | 8163.4986 (71.7)
  AUC (0-24); Day 14; n=9 | 9941.5681 (53.5)
  AUC(0-inf); Day 1; n=7: number analyzed (Participants) | 7
  AUC(0-inf); Day 1; n=7 | 10162.0636 (66.1)
  AUC(0-inf);Day 14; n=7: number analyzed (Participants) | 7
  AUC(0-inf);Day 14; n=7 | 13798.7637 (66.7)
  AUC (0-t); Day 1; n=9 | 7506.5587 (72.3)
  AUC (0-t); Day 14; n=9 | 11861.0783 (59.5)
Statistical Analysis 1: Comparison: 2000 µg OD; Test type: Other; Ratio = 1.22, 90% CI 2-sided [1.01 to 1.47], Standard Error of Mean 0.098 — Treatment ratio of adjusted geometric mean (Day 14/Day 1) for AUC(0-24) is presented

23. Secondary Outcome: Part A: Maximum Observed Plasma Drug Concentration (Cmax) of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Five min post dose concentrations on Days 2-13 were assumed to be the Cmax values. Data for Cmax of GSK2292767 for part A is presented. Cmax is defined as maximum observed plasma concentration of GSK2292767.
Time Frame: Pre-dose (5 min, 30 min, 45 min, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr post dose in each of the 3 treatment periods
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 9 | 12
Picograms per milliliter | 36.9018 (31.9) | 90.8927 (30.6) | 170.7836 (43.7) | 356.0719 (39.4) | 579.8303 (39.5) | 1325.3877 (44.9)
Statistical Analysis 1: Comparison: 50 µg OD vs 100 µg OD; Test type: Other; ratio = 0.78, 90% CI 2-sided [0.61 to 0.99], Standard Error of Mean 0.145
Statistical Analysis 2: Comparison: 100 µg OD vs 200 µg OD; Test type: Other; ratio = 0.96, 90% CI 2-sided [0.75 to 1.22], Standard Error of Mean 0.145
Statistical Analysis 3: Comparison: 100 µg OD vs 500 µg OD; Test type: Other; ratio = 0.81, 90% CI 2-sided [0.68 to 0.97], Standard Error of Mean 0.106
Statistical Analysis 4: Comparison: 100 µg OD vs 1000 µg OD; Test type: Other; ratio = 0.66, 90% CI 2-sided [0.51 to 0.86], Standard Error of Mean 0.154
Statistical Analysis 5: Comparison: 100 µg OD vs 2000 µg OD; Test type: Other; ratio = 0.76, 90% CI 2-sided [0.63 to 0.90], Standard Error of Mean 0.106

24. Secondary Outcome: Part B: Cmax of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Five minute post dose concentrations on Days 2-13 were assumed to be the Cmax values. Data for Cmax of GSK2292767 for part B is presented.
Time Frame: as for outcome 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | 2000 µg OD
Number analyzed (Participants) | 9
Picograms per milliliter
  Day 1 | 1145.7369 (45.9)
  Day 2 | 804.0363 (40.9)
  Day 3 | 871.6343 (38.0)
  Day 4 | 836.4375 (36.0)
  Day 5 | 764.7799 (35.5)
  Day 6 | 785.9632 (49.0)
  Day 7 | 877.1960 (37.7)
  Day 8 | 780.2829 (42.0)
  Day 9 | 745.6613 (35.2)
  Day 10 | 829.2395 (41.8)
  Day 11 | 952.5536 (40.1)
  Day 12 | 881.2328 (46.0)
  Day 13 | 888.9151 (42.9)
  Day 14 | 1305.8068 (41.9)
Statistical Analysis 1: Comparison: 2000 µg OD; Test type: Other; ratio = 1.14, 90% CI 2-sided [0.96 to 1.36], Standard Error of Mean 0.104 — Treatment ratio of adjusted geometric mean (Day 14/Day 1) for Cmax is presented

25. Secondary Outcome: Part A: Time to Maximum Observed Plasma Drug Concentration (Tmax) of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Data for Tmax of GSK2292767 for part A is presented.
Time Frame: as for outcome 23
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 9 | 12
Hours | 1.0046 [0.083 to 3.006] | 0.7540 [0.086 to 4.002] | 0.7500 [0.085 to 3.006] | 0.7583 [0.085 to 4.001] | 1.0264 [0.509 to 2.000] | 1.0125 [0.502 to 3.010]

26. Secondary Outcome: Part B: Tmax of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Data for Tmax of GSK2292767 for part B is presented.
Time Frame: as for outcome 22
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | 2000 µg OD
Number analyzed (Participants) | 9
Hours
  Day 1 | 1.0056 [0.083 to 4.004]
  Day 14 | 1.0050 [0.085 to 3.008]

27. Secondary Outcome: Part A: Terminal Half-life (T1/2) of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Data for T1/2 of GSK2292767 for part A is presented. T1/2 is defined as the time required for one half of the total amount of a particular substance in a biological system to be degraded by biological processes. Only those participants with data available at the specified time points were analyzed.
Time Frame: as for outcome 23
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 0 | 2 | 5 | 7 | 6 | 10
Hours |  | 1.6658 (32.1) | 2.3157 (16.9) | 3.9789 (57.6) | 3.1712 (30.2) | 6.3179 (35.8)

28. Secondary Outcome: Part B: T1/2 of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Data for T1/2 of GSK2292767 for part B is presented. T1/2 was defined as the time required for one half of the total amount of a particular substance in a biological system to be degraded by biological processes. Only those participants with data available at the specified time points were analyzed.
Time Frame: as for outcome 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 2000 µg OD
Number analyzed (Participants) | 7
Hours
  Day 1 | 6.4625 (35.0)
  Day 14 | 11.7665 (48.6)

29. Secondary Outcome: Part A: Trough Concentrations (Ctau) of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Data for Ctau of GSK2292767 for part A is presented. Ctau is defined as the lowest concentration reached by a drug before the next dose is administered.
Time Frame: 24 hr post dose in each of the 3 treatment periods
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | 50 µg OD | 100 µg OD | 200 µg OD | 500 µg OD | 1000 µg OD | 2000 µg OD
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 3 | 11
Picograms per milliliter |  |  |  | 43.5566 (65.9) | 44.1985 (46.4) | 71.6727 (55.6)

30. Secondary Outcome: Part B: Ctau of GSK2292767
Description: Blood samples were collected for pharmacokinetic analysis of GSK2292767 at the specified time points. Data for Ctau of GSK2292767 for part B is presented. Ctau is defined as the lowest concentration reached by a drug before the next dose is administered. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Pico grams per milliliter
Arm/Group | 2000 µg OD
Number analyzed (Participants) | 9
Pico grams per milliliter
  Day 1;n=8: number analyzed (Participants) | 8
  Day 1;n=8 | 78.4862 (91.4)
  Day 2;n=9 | 103.4247 (83.8)
  Day 3;n=9 | 98.3515 (84.1)
  Day 4;n=9 | 112.5132 (83.4)
  Day 5;n=9 | 98.4430 (87.6)
  Day 6;n=9 | 106.6896 (96.2)
  Day 7;n=9 | 101.1219 (88.3)
  Day 8;n=8: number analyzed (Participants) | 8
  Day 8;n=8 | 116.9160 (62.4)
  Day 9;n=9 | 105.3676 (81.7)
  Day 10;n=9 | 117.8348 (80.5)
  Day 11;n=9 | 112.3146 (66.4)
  Day 12;n=8: number analyzed (Participants) | 8
  Day 12;n=8 | 129.6370 (62.8)
  Day 13;n=8: number analyzed (Participants) | 8
  Day 13;n=8 | 154.5480 (52.6)
  Day 14;n=9 | 138.2161 (96.7)
Statistical Analysis 1: Comparison: 2000 µg OD; Test type: Other; Ratio = 2.06, 90% CI 2-sided [1.67 to 2.55], Standard Error of Mean 0.128 — Treatment ratio of adjusted geometric mean (Day 14/Day 1) for Ctau is presented

31. Secondary Outcome: Part B: Concentration of GSK2292767 in Bronchoalveolar Lavage (BAL)
Description: BAL samples were collected by bronchoscopy.
Time Frame: Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | 2000 µg OD
Number analyzed (Participants) | 8
Picograms per milliliter | 8852.94 (236.8)

32. Secondary Outcome: Part B: Concentration of GSK2292767 in Lung Epithelial Lining Fluid (ELF)
Description: ELF from the lung was extracted from BAL samples. ELF drug concentration was calculated as BAL fluid drug concentration multiplied by dilution factor where dilution factor = Plasma urea (pre-bronchoscopy) divided by BAL urea. NA indicates data not available. Only participants with data available at specified time points were analyzed (represented by n=X in category titles).
Time Frame: Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliters
Arm/Group | 2000 µg OD
Number analyzed (Participants) | 9
Picograms per milliliters
  24 Hr Wash 1,n=0: number analyzed (Participants) | 0
  24 Hr Wash 2,n=8: number analyzed (Participants) | 8
  24 Hr Wash 2,n=8 | 9777.25 (290.8)
  24 Hr Wash 3,n=7: number analyzed (Participants) | 7
  24 Hr Wash 3,n=7 | 11921.13 (251.4)

ADVERSE EVENTS:
Time Frame: nSAEs and SAEs were collected from start of study treatment up to 16 weeks
Description: nSAEs and SAEs were collected in Safety Population
Groups:
- Part A: Placebo: Participants administered a single dose of placebo using ELLIPTA DPI via inhalation route.
- Part A: 50 µg OD: Participants administered a single dose of 50 µg GSK2292767 via inhalation route using ELLIPTA DPI
- Part A: 100 µg OD: Participants administered a single dose of 100 µg GSK2292767 via inhalation route using ELLIPTA DPI
- Part A: 200 µg OD: Participants administered a single dose of 200 µg GSK2292767 via inhalation route using ELLIPTA DPI
- Part A: 500 µg OD: Participants administered a single dose of 500 µg GSK2292767 via inhalation route using ELLIPTA DPI
- Part A: 1000 µg OD: Participants administered a single dose of 1000 µg GSK2292767 via inhalation route using ELLIPTA DPI
- Part A: 2000 µg OD: Participants administered a single dose of 2000 µg GSK2292767 via inhalation route using ELLIPTA DPI
- Part B: 2000ug OD: Participants were administered 2000 µg GSK2292767 once daily for 14 days via inhalation route using ELLIPTA DPI
Arm/Group | Part A: Placebo | Part A: 50 µg OD | Part A: 100 µg OD | Part A: 200 µg OD | Part A: 500 µg OD | Part A: 1000 µg OD | Part A: 2000 µg OD | Part B: Placebo | Part B: 2000ug OD
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/12 | 0/12 | 0/13 | 0/12 | 0/9 | 0/12 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/12 | 0/12 | 0/13 | 0/12 | 0/9 | 0/12 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 6/23 | 9/12 | 6/12 | 7/13 | 6/12 | 4/9 | 5/12 | 3/3 | 8/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=23) | Part A: 50 µg OD (N=12) | Part A: 100 µg OD (N=12) | Part A: 200 µg OD (N=13) | Part A: 500 µg OD (N=12) | Part A: 1000 µg OD (N=9) | Part A: 2000 µg OD (N=12) | Part B: Placebo (N=3) | Part B: 2000ug OD (N=9)
Rhythm idioventricular (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 4 | 2 | 1 | 2 | 2 | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchoscopy abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Sputum abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT03045887/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT03045887/SAP_001.pdf